CLINICAL TRIAL: NCT00781404
Title: Myocardial Protection During reperfusión in Patients With Acute Coronary Syndrome With ST Segment Elevation Submitted to Primary Angioplasty: Effect of Intracoronary Adenosine on Infarct Size and Ventricular Remodeling.
Brief Title: Myocardial Protection With Adenosine During Primary Percutaneous Coronary Intervention in Pts With STEMI
Acronym: PROMISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: David Garcia-Dorado (Other)
Collaborators: Hospital General Universitario Gregorio Marañon (Other); Hospital Clínico Universitario de Valladolid (Other); Hospital Universitario Virgen Macarena (Other); Instituto de Ciencias del Corazon (Other)
Responsible Party: Sponsor-Investigator, David Garcia-Dorado, MD, Hospital Universitari Vall d'Hebron Research Institute
Organization: Hospital Universitari Vall d'Hebron Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUValldHebronRI; 2007-006671-36 (EudraCT Number)
Record Dates: First submitted 2008-10-28; First posted 2008-10-29 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Acute Myocardial Infarction
Keywords: adenosine; angioplasty; acute myocardial infarction; acute coronary syndrome with ST segment elevation; infarct size; rescued myocardium
MeSH Terms: interventions — Adenosine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Adenosine — Single dose of adenosine. Solution for infusion of 0.45 mg/mL. Enteral use.
  Other Names: Adenocor

SUMMARY:
OBJECTIVE: to evaluate the safety and efficacy of a brief intracoronary infusion of ADO applied at the time of reperfusion to limit infarct size and LV remodelling in patients with ACSST submitted to primary ACTP.

DESIGN: Multicentric, prospective, randomised, parallel, placebo-controlled double-blind study.

PATIENTS: 200 patients older than 18 with ACSST and without prior myocardial infarction receiving primary PTCA within 6 hours after symptom onset.

DETAILED DESCRIPTION:
The main mechanism responsible for the sanitary impact of ischemic heart disease is cardiomyocyte cell death associated to acute coronary syndrome with ST segment elevation (ACSST). In most of these patients, performing PTCA or thrombolysis as soon as possible does not prevent the occurrence of myocardial necrosis involving a substantial portion of the area at risk. Intracoronary adenosine (ADO) at the time of reperfusion limits infarct size in animals, and preliminary clinical studies indicate that may be also protective in patients with ACSST receiving early reperfusion therapy. OBJECTIVE: to evaluate the safety and efficacy of a brief intracoronary infusion of ADO applied at the time of reperfusion to limit infarct size and LV remodelling in patients with ACSST submitted to primary ACTP. DESIGN: Multicentric, prospective, randomised, parallel, placebo-controlled double-blind study. PATIENTS: 200 patients older than 18 with ACSST and without prior myocardial infarction receiving primary PTCA within 6 hours after symptom onset. PROTOCOL: Intracoronary ADO (4mg) or placebo (saline) infusion distal to the culprit lesion immediately before stent deployment, NMR between 6 and 14 days and after 6 months. END-POINTS: Major: infarct size as measured by NMR, Secondary: changes in LV volumes and EF, and major cardiac events during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years.
* patients with acute coronary syndrome with ST segment elevation within six hours of the onset of symptoms.

Exclusion Criteria:

* patients younger than 18 years and pregnant women.
* patients with previous transmural infarction.
* patients with clinical evidence of bronchospastic lung disease or prior bronchodilator therapy.
* patients with pacemakers.
* patients with TIMI flow higher than 1 and lower than 3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2008-10; Primary Completion 2012-05 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Infarct size measured by MRI | between 5 and 10 days after acute myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: David García-Dorado, MD, PhD, Principal Investigator — Valle Hebron Hospital
Locations (1):
- ValldHebron Hospital, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Garcia-Dorado D, Garcia-del-Blanco B, Otaegui I, Rodriguez-Palomares J, Pineda V, Gimeno F, Ruiz-Salmeron R, Elizaga J, Evangelista A, Fernandez-Aviles F, San-Roman A, Ferreira-Gonzalez I. Intracoronary injection of adenosine before reperfusion in patients with ST-segment elevation myocardial infarction: a randomized controlled clinical trial. Int J Cardiol. 2014 Dec 20;177(3):935-41. doi: 10.1016/j.ijcard.2014.09.203. Epub 2014 Oct 7. PMID 25449504